CLINICAL TRIAL: NCT03522467
Title: Cannabis Oil for Pain Effectiveness
Acronym: COPE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aurora Cannabis Inc (Industry)
Collaborators: Ontario Clinical Oncology Group (OCOG) (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2017-COPE
Record Dates: First submitted 2018-04-27; First posted 2018-05-11 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Cancer; Chronic Pain
Keywords: Cannabis oil; Cannabis; Pain; Cancer
MeSH Terms: conditions — Neoplasms; Chronic Pain; Marijuana Abuse; Pain | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRCP001 (Experimental): MRCP001 administered per protocol dose titration regimen (beginning at 1 capsule daily, titrated to a maximum of 3 capsules BID)
  Interventions: Drug: MRCP001

INTERVENTIONS:
Drug: MRCP001 — MRCP001 is a formulated whole-plant cannabis oil extract, that may help manage poorly controlled chronic pain.
  Other Names: Cannabis oil capsule

SUMMARY:
This project represents a first systematic, prospective, single-arm cohort study of a safe and effective dosing regimen of an orally administered cannabis oil formulation in a cancer subject population with poorly controlled pain.

DETAILED DESCRIPTION:
Over a 1-2 year period, 40 cancer patients experiencing poorly controlled pain will be enrolled in to a prospective single-arm cohort study, in which they will receive an orally administered cannabis oil formulation as an add-on therapy to current treatment regimens. Subjects entering the acute study phase will be titrated to a tolerated dose at which a sustained pain response is reached, and may subsequently enter a 12 week chronic phase during which safety and durability of pain response will be assessed at their stable dose.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with breast, prostate, lung, gastrointestinal or genitourinary cancer who have poorly controlled pain defined by the use of three or more PRN, or as needed, doses of opioids in a 24-hour period for a minimum of three days per week in the week prior to study registration.
2. Age 25-70 years.
3. An ESAS score of 2 or more recorded as their worst pain at the time of study registration.

Exclusion Criteria:

1. Current use of cannabis within the last 30 days from date of study consent (urine screen test positive).
2. Brain metastases.
3. ECOG performance > 2.
4. Life expectancy < 6 months.
5. Daily morphine milligram equivalent (MME) dose < 15 or > 120.
6. Current major psychiatric illness, such as bipolar disorder, major depression, active suicidal intent or psychosis that could be exacerbated by the administration of cannabis.
7. Chemotherapy induced neuropathy.
8. Poorly controlled hypertension, unstable angina, or myocardial infarction within the previous 6 months.
9. Known history or presence of any clinically significant hepatic, renal/genitourinary, gastrointestinal, cardiovascular (e.g. arrhythmias, ischemic heart disease, tachycardia), cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric (e.g. depression, disorientation, euphoric mood and dissociation), dermatological or hematological disease or condition unless determined as not clinically significant.
10. Women who are not practicing an effective form of birth control (condoms, diaphragm, birth control pill, IUD) or are currently pregnant or lactating.
11. Anticipated change in chemotherapy or radiotherapy treatment plan during the 43-day course of the acute study.
12. Known history of substance abuse.
13. Inability to speak or read English.
14. Inability to provide informed consent.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-25 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Sustained pain response | 43 days (Acute Phase)
  Two successive pain responses (Reduction in pain as measured by the Brief Pain Inventory - Short form (BPI-SF) with no increase MME or decrease in MME, continuing for 7 days after dose stabilization)

SECONDARY OUTCOMES:
Pain response at any time | 43 days (Acute Phase) + 12 weeks (Chronic Phase)
  Reduction in pain as measured by the BPI-SF with no increase MME or decrease in MME
Toxicity of treatment intervention - incidence and grade of AEs | 43 days (Acute Phase) + 12 weeks (Chronic Phase)
  As measured by NCIC CTE
Anxiety and depression | 43 days (Acute Phase) + 12 weeks (Chronic Phase)
  As measured by the Hospital Anxiety and Depression Scale (HADS) in which 14 questions are scored on a scale of 0-3. A cumulative score of ≥ 11 will result in a subject being classified as having anxiety and depression using the HADS anxiety and depression, respectively.
Functional well-being | 43 days (Acute Phase) + 12 weeks (Chronic Phase)
  As measured by the Edmonton Symptom Assessment Scale (ESAS), which is routinely performed in most cancer centres in Ontario, and scores pain as well as other cancer-related symptoms between 0-10, 10 being worst possible.
Quality of life change | 43 days (Acute Phase) + 12 weeks (Chronic Phase)
  As measured by the Functional Assessment of Cancer Therapy (FACT-G)
Neuropathic pain | 43 days (Acute Phase) + 12 weeks (Chronic Phase)
  As measured by the Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS), a scale which assigns scores between 0-5 to 7 pain-related outcomes, a cut off ≥ 12 classifying subjects as predominantly having neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Slaven, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No